CLINICAL TRIAL: NCT07217509
Title: PPDTM CorEvitasTM Myasthenia Gravis (MG) Drug Safety and Effectiveness Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-MGR-720
Record Dates: First submitted 2025-09-08; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The design is a prospective, observational (non-interventional) registry for subjects with myasthenia gravis under the care of a neurology provider. Longitudinal data are collected from both subjects and their treating neurology provider during routine clinical encounters using a structured and standardized data collection method. Approximately 1,500 myasthenia gravis subjects with no defined upper limit and 50 clinical neurology sites will be recruited.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of myasthenia gravis subjects to evaluate long-term real-world safety and effectiveness of standard of care treatments for myasthenia gravis. Data collected through the registry may be used to address a range of research questions and use cases, including but not limited to: characterizing the natural history of the disease, evaluating the effectiveness and safety of commercially available medications for the treatment of myasthenia gravis, providing information to support ongoing risk-benefit evaluation by drug manufacturers and regulators, and research related to drug utilization, disease burden, and unmet needs. Further, data collected will inform clinical decision making by patients and treating providers.This provides an opportunity to evaluate other aspects of the disease and its treatment including but not limited to clinical and drug cost-effectiveness, health care resource utilization, and subject adherence

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this registry, an individual must meet all the following criteria:

  1. Has been diagnosed with myasthenia gravis by a neurologist or a qualified neurology practitioner.
  2. Is at least 18 years of age or older and has attained the legal age for consent to procedures involved in the research, under the applicable law of the jurisdiction in which the research is being conducted at the time of enrollment.
  3. Willing and able to provide informed consent.
  4. Willing and able to provide Personally Identifiable Information (full legal name, sex at birth, date of birth, home address zip/postal code and email address or phone Number at a minimum) if required based on registry location and applicable laws and regulations.
  5. In addition, subject must meet at least one of the criteria:

     1. Have started taking a new Enrollment Eligible Medication within 12 months prior to the Enrollment visit. A new medication is a medication that the subject has never taken before.

        OR
     2. Is initiating (prescribed or starting) a new Enrollment Eligible Medication at the Enrollment visit. A new medication is a medication that the subject has never taken before.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in the registry:

  1. Is participating or planning to participate in a double-blind clinical trial for a myasthenia gravis drug. Note: Concurrent participation in another observational registry or open-label Phase 3b/4 trial is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are enrolled in the MG Registry during regularly scheduled office visits. Selected neurologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
MG epidemiology | Every 6 months for 10 years
  The major clinical outcome include an assessment of the epidemiology of Myasthenia Gravis; to better understand the presentation and natural history. This will be determined using PROs and ClinROs which will be included as part of the case report forms.

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No